CLINICAL TRIAL: NCT00002832
Title: Phase I/II Trial of Decitabine and Allogeneic Peripheral Blood Stem Cells Transplantation for Treatment of Relapse Post Allogeneic Bone Marrow Transplantation
Brief Title: Decitabine and Peripheral Stem Cell Transplantation in Treating Patients Who Have Relapsed Following Bone Marrow Transplantation for Leukemia, Myelodysplastic Syndrome, or Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM94-077; P30CA016672 (NIH); MDA-DM-94077 (Other: UT MD Anderson Cancer Center); NCI-G96-1000; CDR0000065034 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: Decitabine; Dacogen; Filgrastim; G-CSF; Neupogen; Cyclosporine; Sandimmune; CYA; Cyclosporin A; Peripheral blood stem cells; PBSC; Allogeneic bone marrow transplantation; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; previously treated myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Blast Crisis | interventions — Filgrastim; Cyclosporine; Decitabine; Stem Cell Transplantation; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decitabine + Stem Cell Transplantation (Experimental)
  Interventions: Biological: Filgrastim; Drug: Cyclosporine; Drug: Decitabine; Procedure: Allogeneic Bone Marrow Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: Filgrastim — Subcutaneously (SQ) daily every 12 hours starting 2-4 days prior to first PBSC collection then daily starting 1 day after PBSC infusion until blood counts recover.
  Other Names: C-CSF; Neupogen
Drug: Cyclosporine — IV daily on day -2, then orally once dose is tolerable, dose may be escalated.
  Other Names: Sandimmune; CYA; Cyclosporin A
Drug: Decitabine — IV for 6 hours every 12 hr for 5 days.
  Other Names: Dacogen
Procedure: Allogeneic Bone Marrow Transplantation — Stem cell infusion on Day 0.
  Other Names: ASCT; Stem Cell Transplantation
Procedure: Peripheral Blood Stem Cell Transplantation — Peripheral blood stem cells (PBSC) are administered 5 days after last dose of decitabine.
  Other Names: PBSC

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be an effective treatment for leukemia, myelodysplastic syndrome, or chronic myelogenous leukemia that has relapsed following bone marrow transplantation.

PURPOSE: Phase I/II trial to study the effectiveness of decitabine and peripheral stem cell transplantation in treating patients who have leukemia, myelodysplastic syndrome, or chronic myelogenous leukemia that has relapsed after bone marrow transplantation.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of decitabine in patients with relapse post allogenic bone marrow transplant. II. Determine the toxicity of decitabine combined with filgrastim (G-CSF) primed allogeneic peripheral blood stem cells in patients who relapsed within 1 year after allogeneic bone marrow transplantation. III. Determine the effectiveness in reinducing remission in these patients.

OUTLINE: Patients receive decitabine IV for 6 hours every 12 hr for 5 days. Peripheral blood stem cells (PBSC) are administered 5 days after last dose of decitabine. Donors receive filgrastim subcutaneously (SQ) daily every 12 hours starting 2-4 days prior to first PBSC collection. If insufficient number of cells are collected, bone marrow can be harvested for supplementation. Donor cells should be collected prior to decitabine infusion. Patients receive filgrastim SQ administered daily starting 1 day after PBSC infusion until blood counts recover. For GVHD prophylaxis, patients receive cyclosporine IV daily on day -2, then orally once dose is tolerable. Dose of decitabine is escalated in cohorts of 3-6 patients. If dose limiting toxicity occurs in 2 of 6 patients at a given dose level, then that dose is declared the maximum tolerated dose. Patients are followed weekly. If none of the first 5 patients survive in remission for more than 100 days, the study will be terminated.

PROJECTED ACCRUAL: At least 15 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute leukemia, myelodysplastic syndromes or chronic myelogenous leukemia (CML) in accelerated phase or blast crisis and relapsed within 1 year after allogeneic bone marrow transplantation Must not be candidates for second course of high dose chemoradiotherapy

PATIENT CHARACTERISTICS: Age: 60 and under Performance status: Zubrod 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 3 mg/dL Renal: Creatinine less than 2 mg/dL Cardiovascular: Greater than 40% ejection fraction per MUGA scan or ECHO Other: Not pregnant No serious intercurrent illness No active CNS disease Must be ineligible for protocols of higher priority No active acute graft vs host disease (GVHD) greater than grade 2 or extensive chronic GVHD No active uncontrolled infection Original marrow donor must undergo filgrastim primed peripheral blood stem cell collection

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 1995-08; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) Decitabine | Weekly for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Giralt, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org